CLINICAL TRIAL: NCT03374332
Title: Fractionated Gemtuzumab Ozogamicin Followed by Non-engraftment Donor Leukocyte Infusions for Relapsed/Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 345
Record Dates: First submitted 2017-11-29; First posted 2017-12-15 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Refractory; progression; recurrence
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Disease Progression; Recurrence | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment 1: Gemtuzumab Ozogamicin and DLI Dose Level 1 (Experimental): Patients ≥70 years old: GO 6mg/m2 (2mg/m2 each dose)
  Patients < 70 years old: GO 9mg/m2 (3mg/m2 each dose)
  Day 8: The product will be administered unprocessed on day 8 (same day as leukapheresis) with a minimum of 1x10^7 CD3+ cells and maximum of 2x10^7 CD3+ cells/kg irrespective of the number of CD34+ cells.
  Patients who show a transient response to therapy can receive up to two additional donor leukocyte infusions with GO 6mg/m2 (2mg/m2 each day, capped at 4.5mg) for all patients regardless of age administered on days 1,4, and 7, no sooner than 35 days status post their last cellular infusion.
  Interventions: Drug: Gemtuzumab Ozogamicin (GO); Other: Donor Leukocytes
- Treatment 2: Gemtuzumab Ozogamicin and DLI Dose Level 2 (Experimental): Patients ≥70 years old: GO 6mg/m2 (2mg/m2 each dose)
  Patients: < 70 years old: GO 9mg/m2 (3mg/m2 each dose)
  Day 8: The product will be administered unprocessed on day 8 (same day as leukapheresis) with a minimum of 1x10^8 CD3+ cells and maximum of 2x10^8 CD3+ cells/kg irrespective of the number of CD34+ cells.
  Patients who show a transient response to therapy can receive up to two additional donor leukocyte infusions with GO 6mg/m2 (2mg/m2 each day, capped at 4.5mg) for all patients regardless of age administered on days 1,4, and 7, no sooner than 35 days status post their last cellular infusion.
  Interventions: Drug: Gemtuzumab Ozogamicin (GO); Other: Donor Leukocytes

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin (GO) — Patients will be given gemtuzumab ozogamicin on days 1,4, and 7. Capped at 4.5mg individual doses. Total doses capped at 13.5mg.
  Other Names: Mylotarg
Other: Donor Leukocytes — The product will be administered unprocessed on day 8/24 hours post GO (same day as leukapheresis) with a minimum of CD3+ cells and maximum of CD3+ cells/kg irrespective of the number of CD34+ cells.

SUMMARY:
This study includes patients with relapsed acute leukemia who have previously been treated with standard treatment that is still present and there is no curative treatment option available. Researchers are studying whether the drug Gemtuzumab Ozogamicin, followed by an infusion of blood cells called leukocytes from a donor, can stimulate the immune system to potentially fight the leukemia. Gemtuzmab ozogamicin is a class of drugs known as an antibody drug conjugate. The drug is given on days 1,4,7. It is infused, attaches to cells with a certain marker on the surface (the majority of which would be leukemia cells). The drug is then internalized and the chemotherapy drug becomes activated. Gemtuzumab is currently FDA approved for the treatment of acute myeloid leukemia.

The infusion of leukocytes to stimulate the immune system to fight your leukemia is investigational and has not been proven to cure cancer. This combination of Gemtuzumab Ozogamicin and donor leukocytes is not an FDA approved treatment and is investigational.

Initially a total of 6 patients will be included in the study to assess the safety of the treatment. Once 6 patients have been treated and no unacceptable toxicities are seen, more patients will be enrolled. The study will treat up to 18 patients on the study.

ELIGIBILITY:
Inclusion Criteria of Recipient (patient):

* Histologic confirmation of acute myeloid leukemia (AML)
* Recurrence or progression (including refractory disease) of AML after at least 1 prior standard treatment with progression within 6 months from last treatment.
* No curative treatment option is available
* ≥ 4-weeks since prior chemotherapy or radiation to cellular therapy infusion.
* Age equal to or greater than 18 years.
* Patients with a history of invasive second malignancy who are disease free for ≥ 2 years.
* Patients must have an expected life expectancy of at least 2 months at the time of initiation of treatment
* No active systemic infections allowed.
* Patients who have relapsed after standard autologous stem cell infusion are eligible as long as they meet all inclusion criteria and no exclusion criteria. These patients must be out more than 6 months from cell infusion to be eligible for enrollment.
* DLCO ≥ 40% with no symptomatic pulmonary disease.
* LVEF ≥ 40% by MUGA or echocardiogram.
* Creatinine <1.5x ULN or any serum creatinine level associated with a measured or calculated creatinine clearance of >40 mL/min, AST and ALT < 2.5x ULN, Total Bilirubin < 1.5 x ULN
* Women of childbearing potential and sexually active males must use 2 forms of effective contraception method from time of consent through 6 months after completing treatment (whether last treatment is infusion or drug).
* Not pregnant or nursing. Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to beginning of treatment (drug). Post-menopausal women (surgical menopause or lack of menses ≥12 months) do not need to have a pregnancy test, please document status.
* Performance status ≤ 2 (or KPS 70)

Exclusion Criteria of Recipient (patient):

* Evidence of HIV infection.
* Any uncontrolled severe, concurrent illness which in the opinion of the treating physician would make this protocol treatment unreasonably hazardous for the patient.
* Oxygen dependent obstructive pulmonary disease.
* Failure to demonstrate adequate compliance with medical therapy and follow-up
* Significant medical or psychiatric illness that would impair the ability to participate in protocol therapy.
* Previous allogeneic stem cell transplant
* Patients who have had previous purine analog (fludarabine, pentostatin, 2-CDA) treatment or treatment with alemtuzumab within 1 year of entering the study
* Previous history of Veno-occlusive disease/Sinusoidal Obstruction Syndrome
* Active hepatitis B or C
* Patients with known active central nervous system leukemia
* Patients with prior treatment of Gemtuzumab ozogamicin
* Patients eligible for allogeneic stem cell transplant

Donor Eligibility Criteria * donor eligibility must be documented and assessed by a separate participating physician other than the treating physician of the recipient.

* Donors agree to up to 3 donor leukocyte collections as documented by assessing physician (although it is not required that the same donor is used for all leukocyte infusions it is preferable, therefore agreement is important at screening). This must be documented in writing by treating physician.
* Typing is required at the following loci: HLA A, B, C, and DRB1.
* Patients with a HLA 0/6 to 3/6(using loci A, B, DR) donor match will be able to participate in this protocol.
* Donors must be a first or second degree relative.
* If the patient/recipient is CMV negative, only CMV negative donors are eligible. If the patient/recipient is CMV positive, CMV testing is not required for the donor.
* Although ABO blood type matching is not required given use of apheresis product preference will be made to ABO compatible donors
* Donors must be ≥18 years of age to donate.
* Donor with a history of malignancy other than non-melanoma skin cancers are eligible only if they had a history of a solid tumor malignancy more than five years prior to lymphocyte donation, and are considered to be in longstanding complete remission as documented by a physician. The donor must be healthy and have all testing criteria completed and meet all criteria for stem cell donation.
* The donor will also be assessed by physician who will document behavioral risk for exposure to infectious agents and diseases. Testing will include the following: Human transmissible spongiform encephalopathy, including Creutzfeldt-Jakob disease, communicable disease risks associated with xenotransplantation, Chlamydia trachomatis and for Neisseria gonorrhea, Treponema pallidum (syphilis).This will exclude the donor.
* The donor must be in good general health and not have significant cardiopulmonary, renal, endocrine, or hepatic disease as documented in writing by physician.
* B-HCG urine or serum negative if donor is of childbearing potential within 7 days of PBMC procurement. Not applicable for donors who are Post-menopausal (surgical menopause or lack of menses ≥12 months).
* Donors must have adequate venous access so leukapheresis can be performed via standard peripheral IV without the need for placement of a central venous catheter.

Donor Exclusion Criteria:

* Evidence of infection for HIV-1, HIV-2, syphilis, hepatitis B or C, HTLV 1 or 2, WNV, Chagas.
* Uncontrolled diabetes mellitus. If donor has controlled diabetes this must be documented by physician.
* Active or congestive heart failure syndrome from any cause per donor medical history. Approval for participation by Cardiologist required to be sent to BrUOG.
* Full cardiac workup by a Cardiologist is required for any history of congestive heart failure syndrome, conduction abnormalities or history of arrhythmia other than treated atrial fibrillation.
* Active angina pectoris. To be documented by physician
* Oxygen dependent pulmonary disease. To be documented by physician
* History of any lymphoid, myeloid or other non-solid malignancy. To be documented by physician
* Failure to receive full informed consent.
* Inadequate renal and/or hepatic function per medical history. To be documented by physician
* Known history of cirrhosis or active liver disease per medical history. To be documented by physician
* History of transplantation. To be documented by physician.
* A donor in whom plasma dilution sufficient to affect the results of communicable disease testing is suspected, unless: (A) You test a specimen taken from the donor before transfusion or infusion and up to 7 days before recovery of cells or tissue; or (B) You use an appropriate algorithm designed to evaluate volumes administered in the 48 hours before specimen collection, and the algorithm shows that plasma dilution sufficient to affect the results of communicable disease testing has not occurred.
* Clinical situations in which you must suspect plasma dilution sufficient to affect the results of communicable disease testing will exclude the donor. Such situations include, but are not limited to the following:(A) Blood loss is known or suspected in a donor over 12 years of age, and the donor has received a transfusion or infusion of any of the following, alone or in combination:

  1. More than 2,000 milliliters (mL) of blood (e.g., whole blood, red blood cells) or colloids within 48 hours before death or specimen collection, whichever occurred earlier, or
  2. More than 2,000 mL of crystalloids within 1 hour before death or specimen collection, whichever occurred earlier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Response Rate | Post infusion for a total of 2 years.
  Response rate of infusional gemtuzumab ozogamicin followed by nonengraftment donor leukocyte infusions in patients with refractory acute myeloid leukemia.
  Bone Marrow Biopsy to be done in patients thought to have responded.

SECONDARY OUTCOMES:
Survival | Through 2 years post end of treatment
  Progression free survival and overall survival of infusional gemtuzumab ozogamicin followed by nonengraftment donor leukocyte infusions in patients with refractory acute myeloid leukemia.
Dose limiting toxicities | Start of treatment through 30 days post the final infusion
  Rate of dose limiting toxicities of gemtuzumab ozogamicin followed by nonengraftment donor leukocyte infusions in patients with refractory acute myeloid leukemia.

CONTACTS AND LOCATIONS:
Overall Officials: John Reagan, MD, Principal Investigator — Brown University Oncology Research Group (BrUOG)
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States